CLINICAL TRIAL: NCT07015801
Title: Open-label Individual Patient Study of Cytomegalovirus (CMV)-Specific Donor-derived T Lymphocytes (DTL) for the Treatment of Recalcitrant CMV Infection in a Patient With Primary Immunodeficiency
Brief Title: CMV-specific Donor-derived T Lymphocytes for the Treatment of Recalcitrant CMV Infection in a Patient With Primary Immunodeficiency
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Precision Laboratories (Unknown); Alberta Health services (Other); University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMV-DTL
Record Dates: First submitted 2025-05-22; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Cytomegalovirus Viremia; Cytomegalovirus Pneumonia; T-Lymphocyte Immunodeficiency
Keywords: donor-derived T lymphocytes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CMV-specific donor-derived T lymphocytes (CMV-VST). (Experimental): Mixture of donor lymphocytes, reactive to peptides derived from cytomegalovirus.
  Interventions: Biological: CMV-VST

INTERVENTIONS:
Biological: CMV-VST — 30-40 x 10^3 viable CD3+ cells/kg

SUMMARY:
Treatment of CMV in a patient with profound combined immunodeficiency, who has viremia and pneumonia, using CMV-specific donor-derived T lymphocytes (CMV-VST).

DETAILED DESCRIPTION:
Treatment of CMV in a patient with profound combined immunodeficiency, who has viremia and pneumonia, using CMV-specific donor-derived T lymphocytes (CMV-VST), a cell therapy product containing a mixture of donor lymphocytes, reactive to peptides derived from cytomegalovirus.

After having receipt of therapy, the patient will have clinical assessments twice a week until discharge from the inpatient unit. After discharge, assessments will be performed on a weekly basis for three months. From 3-12 months, the patient will be seen monthly and then every three months till 2 years post planned hematopoietic stem cell transplantation. After 2 years, survival status will be assessed every 6 months through year 15.

ELIGIBILITY:
Inclusion Criteria:

* profound combined immunodeficiency
* cytomegalovirus (CMV) infection
* viremia
* pneumonia

Exclusion Criteria:

* Receiving a steroid dose of ≥ 0.5 mg/kg of prednisolone equivalent
* Receiving antithymocyte globulin or similar anti-T-cell antibody therapy, methotrexate, or other antimetabolite-type immunosuppressants that are toxic to proliferating T cells, and extracorporeal
* Receiving checkpoint inhibitor agents (eg, nivolumab, pembrolizumab, ipilimumab) are within 3 drug half-lives of the most recent dose to cycle 1 day 1.
* Administration of another investigational product

Ages: 0 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2040-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of study | Enrollment to 24 months
  Evaluate the feasibility of conducting this study, evaluated in terms of whether or not the study could be completed as laid out in the protocol in the time allotted.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Weekly to 3 months
  AEs assessed according to CTCAE grading criteria.
Efficacy of Intervention | Weekly to 3 months
  Change in viremia from baseline according to PCR testing after the intervention
Efficacy of Intervention | Monthly from 3 to 12 months
  Change in viremia from baseline according to PCR testing after the intervention
Efficacy of Intervention | Every 3 months from 12-24 months
  Change in viremia from baseline according to PCR testing after the intervention

SECONDARY OUTCOMES:
Engraftment failure | Enrollment to 24 months
  Assessment of evidence of engraftment failure from clinical evaluations
Graft versus host disease | Enrollment to 24 months
  Assessment of evidence of graft versus host disease (GVHD) from clinical evaluations
Transplant associated thrombotic microangiopathy | Enrollment to 24 months
  Assessment of evidence of Transplant associated thrombotic microangiopathy (TA-TMA) from clinical evaluations
Death | Enrollment to 24 months
  Death of participant
CMV-reactive T cell number | Weekly to 3 months
  The number of CMV-reactive T cells in the patient's blood will be enumerated using an CMV-ELISpot assay.
CMV-reactive T cell number | Monthly from 3 to 12 months
  The number of CMV-reactive T cells in the patient's blood will be enumerated using an CMV-ELISpot assay.
CMV-reactive T cell number | Every 3 months from 12-24 months
  The number of CMV-reactive T cells in the patient's blood will be enumerated using an CMV-ELISpot assay.
Total CMV-reactive T cell activity | Weekly to 3 months
  The total amount of INF γ secreted from all CMV-reactive T cells in the patient's blood to measured using a commercially available ELISA kit (QuantiFERON-CMV). This will allow track the cumulative response to CMV by the reactive T cells over time.
Total CMV-reactive T cell activity | Monthly from 3 to 12 months
  The total amount of INF γ secreted from all CMV-reactive T cells in the patient's blood to measured using a commercially available ELISA kit (QuantiFERON-CMV). This will allow track the cumulative response to CMV by the reactive T cells over time.
Total CMV-reactive T cell activity | Every 3 months from 12-24 months
  The total amount of INF γ secreted from all CMV-reactive T cells in the patient's blood to measured using a commercially available ELISA kit (QuantiFERON-CMV). This will allow track the cumulative response to CMV by the reactive T cells over time.
CMV-reactive T cell phenotyping | Weekly to 3 months
  Flow cytometry will be used to characterize CMV-reactive T cell phenotype
CMV-reactive T cell phenotyping | Monthly from 3 to 12 months
  Flow cytometry will be used to characterize CMV-reactive T cell phenotype
CMV-reactive T cell phenotyping | Every 3 months from 12-24 months
  Flow cytometry will be used to characterize CMV-reactive T cell phenotype
RNA sequencing | Weekly to 3 months
  RNA sequencing, to characterize CMV-reactive T cell biology and track individual VST clones
RNA sequencing | Monthly from 3 to 12 months
  RNA sequencing, to characterize CMV-reactive T cell biology and track individual VST clones
RNA sequencing | Every 3 months from 12-24 months
  RNA sequencing, to characterize CMV-reactive T cell biology and track individual VST clones
Serum cytokine analysis | Weekly to 3 months
  Serum cytokines, to estimate total CMV-reactive T cell activity and host response to treatment
Serum cytokine analysis | Monthly from 3 to 12 months
  Serum cytokines, to estimate total CMV-reactive T cell activity and host response to treatment
Serum cytokine analysis | Every 3 months from 12-24 months
  Serum cytokines, to estimate total CMV-reactive T cell activity and host response to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No